CLINICAL TRIAL: NCT01053819
Title: Can We Miss Pigmented Lesions in Psoriasis Patients?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Boni Elewski, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F070629011
Record Dates: First submitted 2009-02-06; First posted 2010-01-21 (Estimated); Results first posted 2012-08-22 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Psoriasis; Melanoma; Non-melanoma Skin Cancer
Keywords: psoriasis; melanoma; non-melanoma skin cancer; etanercept; Enbrel
MeSH Terms: conditions — Psoriasis; Melanoma | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etanercept (Experimental): open label treatment(50 mg SQ)per Food and Drug Administration approval for 24 weeks
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept — Patients will receive six months of treatment with Enbrel 50mg SQ given twice a week for the first three months and 50 mg once a week thereafter.
  Other Names: Enbrel

SUMMARY:
In psoriasis patients, thick psoriatic plaques can obscure these lesions, and clinicians rely heavily on visual inspection to recognize suspicious or atypical pigmented lesions. However, successful systemic treatment and subsequent clearing of psoriatic plaques may allow clinicians to better evaluate pigmented lesions, thereby increasing the likelihood of early identification and treatment of suspicious lesions such as nonmelanoma skin cancer and malignant melanoma.

DETAILED DESCRIPTION:
No further description is desired.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of moderate to severe plaque psoriasis identified by a BSA greater than or equal to 10% and a Psoriasis Area and Severity Index score greater than or equal to 12
2. Age 19 years or above
3. Fitzpatrick skin type I, II or III
4. Candidate for systemic treatment in the opinion of the investigator
5. Willingness to undergo treatment with Enbrel as outlined above
6. Negative pregnancy test (urine or serum β-Human Chorionic Gonadotrophin ) before the first dose of study drug in all women (except those surgically sterile, or at least 5 years postmenopausal).
7. Negative Tuberculosis skin test at entry into the study or a negative screening x-ray in inconclusive Purified Protein Derivative reading (borderline, reactive but non-diagnostic) or in prior bacille Calmette-Guerin inoculated subjects.
8. Sexually active subjects of childbearing potential must agree to use medically acceptable form of contraception during screening and throughout the study
9. Subject or designee must have the ability to self-inject study medication or have a care giver at home who can administer subcutaneous injections
10. Must be able and willing to give written informed consent and comply with the requirements of the study protocol and must authorize release and use of protected health information

Exclusion Criteria:

1. Serum creatinine > 3.0 mg/dL (265 micromoles/L)
2. Serum potassium < 3.5 mmol/L or > 5.5 mmol/L
3. Serum alanine aminotransferase or Aspartate transaminase > 3 times the upper limit of normal for the Lab
4. Platelet count < 100,000/mm3
5. White blood cell count < 3,000 cells/mm3
6. Hemoglobin, hematocrit, or red blood cell count outside 30% of the upper or lower limits of normal for the Lab
7. Systemic therapy use (e.g. phototherapy, methotrexate, cyclosporine, oral steroids, systemic biologics) within the previous 4 weeks
8. Topical therapy use (e.g. topical steroids, vitamin D derivatives) within the previous 2 weeks
9. Subject is currently enrolled in another investigational device or drug trial(s), or subject has received other investigational agent(s) within 28 days of baseline visit.
10. Subjects who have known hypersensitivity to Enbrel or any of its components or who is known to have antibodies to etanercept
11. Prior or concurrent cyclophosphamide therapy
12. Concurrent sulfasalazine therapy
13. Known Human immunodeficiency virus-positive status or known history of any other immunosuppressing disease
14. Active severe infections within 4 weeks before screening visit, or between the screening and baseline visits
15. Untreated Lyme disease
16. Severe comorbidities (diabetes mellitus requiring insulin, CHF of any severity, MI, CVA or TIA within 3 months of screening visit, unstable angina pectoris, uncontrolled hypertension (sitting systolic BP <80 mm Hg or > 160 or diastolic BP > 100 mm Hg), oxygen-dependent severe pulmonary disease, history of cancer within 5 years [other than resected cutaneous basal or squamous cell carcinoma or in situ cervical cancer])
17. History of TB or TB exposure, chronic hepatitis B or hepatitis C, SLE, history of multiple sclerosis, transverse myelitis, optic neuritis or epilepsy
18. History of recent alcohol or substance abuse (< 1 year)
19. Pregnant or lactating females
20. Use of a live vaccine 90 days prior to, or during this study
21. Any condition judged by the patient's physician to cause this clinical trial to be detrimental to the patient
22. History of non-compliance with other therapies

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boni E Elewski, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Dermatology, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Patients will receive six months of treatment with Enbrel 50mg SC given twice a week for the first three months and 50 mg once a week thereafter.
Period: Overall Study
Arm/Group | Etanercept
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Etanercept: open label treatment per FDA approval for 24 weeks
Arm/Group | Etanercept
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint for This Study Will be a Change From Baseline in the Number of Pigmented Lesions on Skin Previously Covered by Psoriatic Plaques.
Time Frame: Patients will complete study within 6 months.
Population: The data for this Outcome was not collected and due to the length of time, the records have been destroyed.
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 6
participants | 0

2. Secondary Outcome: A Secondary Objective Will be to Evaluate the Identified Pigmented Lesions for Suspicious Criteria
Description: The data for this Outcome was not collected and due to the length of time, the records have been destroyed.
Time Frame: Patients will complete the study within 6 months
Population: The data for this Outcome was not collected and due to the length of time, the records have been destroyed.
Arm/Group | Etanercept
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes